CLINICAL TRIAL: NCT05128708
Title: Safety and Feasibility of the Combined Medial and Caudal Approach in Open and Laparoscopic Radical Right Hemicolectomy for Right Colon Cancer
Brief Title: Combined Medial and Caudal Approach for Right Hemicolectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Zakaria Mohamed Ahmed, assistant lecturer of general surgery, Zagazig University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #6199-29-6-2020; zagazig university (Other: faculty of medicine zagazig university)
Record Dates: First submitted 2021-11-04; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Colon Cancer
Keywords: right colon; medial and caudal approach; hemicolectomy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Intervention Model Description: all participants underwent right hemicolectomy using combined medial and caudal approach and divided into 2 groups group I had open surgery and group II had laparoscopic surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open right hemicolectomy (Active Comparator): participants diagnosed as operable right sided colon cancer were enrolled in this study and did open combined medial and caudal resection procedure
  Interventions: Procedure: combined medial and caudal approach right hemicolectomy open and laparoscopic
- laparoscopic right hemicolectomy (Active Comparator): participants diagnosed as operable right sided colon cancer were enrolled in this study and did laparoscopic combined medial and caudal resection procedure
  Interventions: Procedure: combined medial and caudal approach right hemicolectomy open and laparoscopic

INTERVENTIONS:
Procedure: combined medial and caudal approach right hemicolectomy open and laparoscopic — resection of right colon cancer by this radical approach

SUMMARY:
Right sided hemicolectomy is the standard type of operation for cancers in the caecum, the ascending colon, proximal transverse colon.The aim of this study was to assess the safety and feasibility of combined medial and caudal approach in performing right hemicolectomy and to compare outcome between laparoscopic and open surgery in right colon cancer.

DETAILED DESCRIPTION:
The incidence of colorectal cancer is increasing. Slight shift towards right colon cancer is noticed in the last 2 decades in Egypt. This can be attributed to advances in diagnostic tools and increased public health awareness as right sided colon cancer was almost presented late as most of tumors located in the capacious cecum. Hence, early diagnosis with good radical procedure offers better outcome, quality of life and survival. Many approaches for right colon resection were described. In this study we adopted the combined medial and caudal approach for right colon resection in cases of right colon cancer in both open and laparoscopic techniques.

Traditionally, approach to right colon cancer is through open exploration but this approach has more blood loss, prolonged postoperative hospital stay, sever postoperative pain and delayed recovery.

As combined medial and caudal approach is a radical procedure,the purpose of the present study was to compare between laparoscopic and open right hemicolectomy both done with combined medial and caudal approach in right colon cancer as regards technical feasibility, advantages and disadvantages of both procedures.

This was prospective randomized study and was carried out on 26 participants as number of cases with right hemicolon cancer is about 2 per month in our center. Those participants diagnosed as operable right sided colon cancer and the participants were divided into two groups:

Group I: Open combined medial and caudal right hemicolectomy included 13 participants Group II: Laparoscopic combined medial and caudal right hemicolectomy included 13 participants

All patients with inclusion criteria were subjected to preoperative assessment in the form of:

* Full history.
* Clinical evaluation.
* Laboratory investigation (Complete blood picture, liver function tests, blood sugar, blood urea, serum creatinine, prothrombin time, serum albumin and tumour marker CEA).
* Imaging (chest X-ray, US abdomen, CT abdomen and pelvis).
* Histopathology diagnosis (endoscopic biopsy, tissue diagnosis).
* Determined whether participants underwent open or laparoscopic operation is multifactorial e.g., patients desire, contraindications for laparoscopy and mass size if more than 5 cm preferred to have open surgery.
* Informed written consent taken from the patients or the legal guardian.

operative technique: both groups offered combined medial and caudal approach

* Fasting for 6 hours with no oral intake or only clear fluids intake the day before or better bowel preparation.
* After confirming the availability of blood of matching blood group, general anesthesia is inducted and prophylactic antibiotics are given.
* Patient positioning:

  1. group I: (Open cases) The standard position for an open right hemicolectomy is supine with strapping of the ankle and wrists, such as the Trendelenburg position. The surgeon stands on the patient's left, and the first assistant stands across from the surgeon on the patient's right. The scrub nurse stands beside the surgeon. If a second assistant is needed, he or she usually stands across from the surgeon to the left of the first assistant.
  2. group II: laparoscopic cases: The patient should be placed in the supine position with his two legs apart and arms tucked beside the body.

The surgeon should stand between the patient's legs with the assistant standing on the patient's left and the camera operator standing on the assistant's left side, and the scrub nurse on the patient's right side.

The video monitor is placed on the patient's upper right.

* Abdominal access and trocar placement by open or closed technique using veress needle for pneumoperitoneum with an intraperitoneal pressure of 14 mmHg.
* The procedure requires 5 trocars.
* A 10 mm trocar is placed 3 cm below umbilicus for the 30° angled telescope to get an adequate view. The incision would be enlarged to extract the specimen and performing anastomosis.
* A12 mm trocar is introduced 5 cm below the telescope port for the surgeon right hand instrument.
* A 5 mm port is inserted at the McBurney's point for the surgeon's left hand instrument.
* Additional two 5 mm trocars are placed at the opposite of McBurney's point and the right subcostal position respectively for the assistant to retract and display the colon and mesocolon.

Intraoperatively, all patients will be assessed for:

* Time of the procedure.
* Amount of blood loss.

post operatively: Postoperative medications given. Monitoring of vital signs and drains. post operative assesment of pain is subjective to the participant as he gave it a score from 1 to 10. minimal pain score(1 to 3), mild (4 to 6) and sever (7 to 10). Ambulation and clear oral fluids started when intestinal sounds are audible followed by soft diet. The intraperitoneal tube drain removed when there is less than 50cc of fluid per 24h or after performing ultrasonography.

Follow up:

Participants are reviewed as outpatients weekly for 1 month or more frequent if they develop any complications between their visits.

The postoperative pathological results, number of lymph node dissection, postoperative exhaust time, postoperative abdominal drain volume and duration, postoperative short term complications, hospital stay and postoperative pathological staging will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed right colon cancer with colonoscopic biopsy.
* No invasion of the surrounding tissue.
* No distant metastasis except the liver.

Exclusion Criteria:

* Informed consent refusal
* Malignancy recurrence
* Distant metastasis except the liver.
* Locally advanced tumor.
* participants need emergent intervention e.g., intestinal obstruction or perforation.
* Contraindications specific for laparoscopy for laparoscopy cases

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
calculate the duration of operation in both groups | The duration of operation was calculated intra operatively from skin incision to skin closure. it was ranging from 2 to 4 hours after skin incision.
  The duration of operation was calculated in minutes in both groups. group I: open combined medial and caudal right hemicolectomy and group II: laparoscopic combined medial and caudal right hemicolectomy from skin incision till skin closure intraoperatively.
Detection of the amount of blood loss during operation in both groups. | the amount of blood loss was detected intra operatively for 4 hours after skin incision.
  the amount of blood loss during operation is calculated in cubic centimetres using scaled container connected to suction device in both groups.
Detection of organ or visceral injury in both groups | detection of organ injury was detected intra operatively for 4 hours after skin incision.
  detection of organ or visceral injury was done intra operatively by naked eye in both groups.
detection of the duration of hospital stay in both groups | duration of hospital stay was detected from the day of operation till the day of discharge (4 to 7 days postoperatively)
  the duration of hospital stay was detected in days in both groups
detection of number of resected lymph nodes in both groups | number of resected lymph nodes was detected from 7th to 10th day post operatively
  the number of resected lymph nodes was detected in post operative histopathological reports in both groups.
detection of occurrence of postoperative pain in both groups | detection of post operative pain in both groups was done from the day of operation to 7 days postoperatively.
  detection of post operative pain was detected in both groups using a written scale fulfilled by the participant giving a score from 1 out of 10 points (1 to 3 points referred as minimal) (4 to 6 points referred as mild) (7 to 10 points referred as sever).
detection of occurrence fecal fistula in both groups | detection of occurrence of fecal fistula in both groups was detected from 2 to 7 days postoperatively
  occurrence of fecal fistula in both groups was detected by vision of fecal discharge in drains from 48 hours post operatively till discharge day.
detection of post operative wound infection in both groups | post operative wound infection in both groups was detected from 2 days to one month post operatively.
  post operative wound infection in both groups was detected by vision of wound discharge or pus.

CONTACTS AND LOCATIONS:
Overall Officials: Reham Z Mohamed, master, Principal Investigator — assistant lecturer of general surgery zagazig university; Ali H Elshewy, PhD, Study Director — professor of general surgery zagazig university; Abdelrahman A Sarhan, PhD, Study Chair — professor of general surgery zagazig university; Gamal M Osman, PhD, Study Director — assistant professor of general surgery zagazig university
Locations (1):
- Zagazig University Hospitals, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No
researchers should contact the principle investigator for individual participant data

REFERENCES:
- [Background] Troisi RJ, Freedman AN, Devesa SS. Incidence of colorectal carcinoma in the U.S.: an update of trends by gender, race, age, subsite, and stage, 1975-1994. Cancer. 1999 Apr 15;85(8):1670-6. PMID 10223559
- [Background] Gouvas N, Agalianos C, Papaparaskeva K, Perrakis A, Hohenberger W, Xynos E. Surgery along the embryological planes for colon cancer: a systematic review of complete mesocolic excision. Int J Colorectal Dis. 2016 Sep;31(9):1577-94. doi: 10.1007/s00384-016-2626-2. Epub 2016 Jul 28. PMID 27469525
- [Background] Jessup JM, McGinnis LS, Steele GD Jr, Menck HR, Winchester DP. The National Cancer Data Base. Report on colon cancer. Cancer. 1996 Aug 15;78(4):918-26. doi: 10.1002/(SICI)1097-0142(19960815)78:43.0.CO;2-W. PMID 8756390
- [Background] Chen Q, Shuai X, Chen L. [Safety and feasibility of the combined medial and caudal approach in laparoscopic D3 lymphadenectomy plus complete mesocolic excision for right hemicolectomy in the treatment of right hemicolon cancer complicated with incomplete ileus]. Zhonghua Wei Chang Wai Ke Za Zhi. 2018 Sep 25;21(9):1039-1044. Chinese. PMID 30269325
- [Background] Li F, Zhou X, Wang B, Guo L, Wang J, Wang W, Fu W. Comparison between different approaches applied in laparoscopic right hemi-colectomy: A systematic review and network meta-analysis. Int J Surg. 2017 Dec;48:74-82. doi: 10.1016/j.ijsu.2017.10.029. Epub 2017 Oct 12. PMID 29032159
- [Background] Xie D, Yu C, Gao C, Osaiweran H, Hu J, Gong J. An Optimal Approach for Laparoscopic D3 Lymphadenectomy Plus Complete Mesocolic Excision (D3+CME) for Right-Sided Colon Cancer. Ann Surg Oncol. 2017 May;24(5):1312-1313. doi: 10.1245/s10434-016-5722-1. Epub 2016 Dec 19. PMID 27995452